CLINICAL TRIAL: NCT06871189
Title: Age and Gender on TMJ Sound Frequencies and Mouth-Opening Distances
Brief Title: Age and Gender in TMJ Sounds
Status: Completed | Type: Observational
Sponsor: Atlas University (Other)
Responsible Party: Principal Investigator, Serdar Gozler, Dr., Atlas University
Other Study IDs: 2024-ATLAS
Record Dates: First submitted 2025-02-28; First posted 2025-03-11 (Actual); Last update posted 2025-03-11 (Actual); Status verified 2025-02

CONDITIONS: Temporomandibular Disorders (TMD)
Keywords: age; gender; temporomandibular disorders; vibration frequencies
MeSH Terms: conditions — Temporomandibular Joint Disorders; Coitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (4):
- Female ≤22 years: Participants who identify as female and are 22 years old or younger.
- Female ≥23 years: Participants who identify as female and are 23 years old or older.
- Male ≤22 years: Participants who identify as male and are 22 years old or younger.
- Male ≥23 years: Participants who identify as male and are 23 years old or older.

SUMMARY:
The temporomandibular joint (TMJ) plays a crucial role in masticatory function, and its proper lubrication is essential for smooth, frictionless movement. Disruptions to the lubricating system, often due to age-related changes or parafunctional activities such as teeth clenching or bruxism, can increase joint friction, leading to vibrations or intra-articular sounds. These sounds have become an essential diagnostic tool for assessing internal derangements of the TMJ. While magnetic resonance imaging (MRI) is considered the gold standard for diagnosing TMJ disorders, its limitations in evaluating intra-articular structures have led to the development of alternative methods, such as Joint Vibration Analysis (JVA). This study explores the relationship between age, gender, and TMJ vibration frequencies using JVA in a cohort of 367 participants. We analyzed four key vibration parameters: Range of Motion (ROM), Total Integral Left (TIL), Total Integral Right (TIR), and frequency distributions in the <300 Hz and >300 Hz segments.

ELIGIBILITY:
Inclusion Criteria:

* Participants capable of achieving an inter-incisal opening of 30 to 50 mm without restrictions.
* Free from symptoms indicative of temporomandibular disorder (TMD).
* Possessing fully and/or prosthetically restored dentition.
* Demonstrating adequate mouth opening to facilitate the rotation of the condylar process.

Exclusion Criteria:

* Individuals using psychotropic or narcotic medications, regardless of medical oversight.
* Regular consumption of painkillers or anti-inflammatory agents.
* Long-term treatment with cortisone or its derivatives. Individuals who have sustained traumatic injuries to the maxillofacial region.
* Participants who have suffered the loss of organs and/or tissue in the maxillofacial area due to medical or traumatic causes.

Ages: 10 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: free of symptoms related to temporomandibular disorder
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2024-12-08 (Actual); Primary Completion 2025-03-05 (Actual); Study Completion 2025-03-05 (Actual)

PRIMARY OUTCOMES:
range of motion | The outcome measure was assessed at baseline.
  ROM is measured as the maximum mouth opening (mouth opening distance), which is an indicator of joint mobility and dysfunction in TMD patients. Limited or abnormal ROM in the TMJ, reflected by restricted mouth opening, is often associated with pain, dysfunction, and impaired jaw movement, making it a crucial parameter for assessing the severity of TMD.
Total Integral | The outcome measure was assessed at baseline
  hese parameters assess the intensity and frequency of the joint's movement on each side (left and right). TIL and TIR represent the overall activity and functional performance of the TMJ during movement, with abnormal values potentially indicating dysfunction or asymmetry between the left and right sides. These parameters are critical for evaluating the joint's response to treatment and the presence of any abnormalities in movement or pressure distribution across the TMJ.
Frequency Components | The outcome measure was assessed at baseline
  The frequency parameters assess the overall movement and condition of the temporomandibular joint (TMJ) by measuring pressure wave activity across different frequency ranges. Integral > 300 Hz (d1/d2) reflects higher frequency components primarily influenced by joint surface roughness and degenerative changes. Integral < 300 Hz (c1/c2) represents lower frequency components associated with disc movements, which can be affected by disc displacement, hypermobility, or joint laxity. The Ratio (e1/e2) indicates the ratio of high to low frequencies, providing insight into joint surface condition and overall TMJ health. These parameters are crucial for evaluating the function and possible degeneration of the TMJ.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Atlas Univercity, Istanbul, Anadolu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol